CLINICAL TRIAL: NCT00158340
Title: Binge Eating Self-Guided Treatment (BEST)
Brief Title: Guided Self-Help Treatment for Binge Eating Disorder
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH066966 (NIH); R01MH066966 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Eating Disorders; Bulimia
Keywords: Binge Eating; Overeating; Compulsive Eating; Hyperphagia
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia; Hyperphagia; Food Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive guided self-help cognitive behavioral therapy
  Interventions: Behavioral: Guided self-help cognitive behavioral therapy (CBT)
- 2 (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Usual clinical care

INTERVENTIONS:
Behavioral: Guided self-help cognitive behavioral therapy (CBT) — Participants receive eight sessions of guided self-help CBT.
  Arms: 1
Behavioral: Usual clinical care — Control group participants receive treatment as usual.
  Arms: 2

SUMMARY:
This study will determine the effectiveness of guided self-help treatment in treating individuals with binge eating disorder (BED).

DETAILED DESCRIPTION:
Binge eating disorder (BED) is a serious condition characterized by compulsive overeating and feelings of powerlessness. The condition often has a negative impact on both physical and emotional health. This study will examine ways to help people determine whether they have BED and will test whether guided self-help (GSH) treatment is effective in treating BED.

Participants will be randomly assigned to receive either GSH treatment or usual clinical care (which may include general support and talk therapy) for 3 months. The GSH treatment is a cognitive behavioral therapy-based program that will be administered over 8 sessions. Participants receiving GSH will be given a book that focuses on dealing with BED; they will also meet with a therapist regularly to have their progress monitored. The Eating Disorders Examination (EDE), self-reports, questionnaires, and surveys will be used to assess participants. Assessments will be conducted at study entry, at Weeks 2 and 4 of the treatment, at the end of the treatment, and at 6 and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of binge eating disorder (BED) bulimia nervosa (BN), or spectrum BN, defined as recurrent binge eating at least once a week for 3 months
* Body mass index (BMI) between 18 and 45
* Continuous membership in the Kaiser Permanente Northwest Division for at least 12 months prior to study entry

Exclusion Criteria:

* Diagnosis of anorexia nervosa or psychotic disorder
* Significant organic brain syndromes, retardation, pervasive developmental disorder, or autism
* At risk for suicide
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2004-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Frequency of binge eating | Measured at post-treatment, Week 12, Month 6, and Year 1

SECONDARY OUTCOMES:
Frequency of inappropriate compensatory behaviors, dietary restraint, over-valuation of weight/shape, functional impairment, self-esteem, and social impairment | Measured at post-treatment, Week 12, Month 6, and Year 1
Body weight | Measured at post-treatmentand Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Ruth H. Striegel-Moore, PhD, Principal Investigator — Wesleyan University
Locations (2):
- United States (2):
  - Wesleyan University Department of Psychology, Middletown, Connecticut
  - Kaiser Permanente Center for Health Research, Portland, Oregon

REFERENCES:
- [Derived] Lynch FL, Striegel-Moore RH, Dickerson JF, Perrin N, Debar L, Wilson GT, Kraemer HC. Cost-effectiveness of guided self-help treatment for recurrent binge eating. J Consult Clin Psychol. 2010 Jun;78(3):322-33. doi: 10.1037/a0018982. PMID 20515208